CLINICAL TRIAL: NCT05030064
Title: Clinical Study on the Efficacy and Safety of Fecal Microbiota Transplantation in the Treatment of Ulcerative Colitis With Depression
Brief Title: Clinical Study on the Fecal Microbiota Transplantation in the Treatment of Ulcerative Colitis With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Yanling Wei, Deputy Chief Physician, Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-DP-GI-FMT-003
Record Dates: First submitted 2021-08-09; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis，Depression，FMT
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Gastrointestinal Microbiome

STUDY DESIGN:
Intervention Model Description: It is planned to recruit UC patients with depression and voluntarily receive standard enterobacteria capsule or placebo treatment. A total of 54 cases will be completely randomized according to the random number table and randomly divided into 2 groups for intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intestinal flora capsule(FMT) (Experimental): The group includes 27patients.They will receive 16 capsules of intestinal bacteria each time, once a week, 4 times in a row.Each capsule contains 200mg of fecal bacteria.
  Interventions: Drug: Intestinal flora capsule
- Placebo group (Placebo Comparator): The group includes 27patients.They will receive 16 Placebo capsules each time, once a week, 4 times in a row.
  Interventions: Procedure: placebo capsule

INTERVENTIONS:
Drug: Intestinal flora capsule — This research group has independently researched and created a human intestinal flora capsule based on "intestinal bacteria transplantation": Intestinal flora capsule, which has been declared a national invention patent (patent number: 2015103040414).
  Other Names: Fecal Bacteria Transplant
  Arms: Intestinal flora capsule(FMT)
Procedure: placebo capsule — Each placebo capsule is the two-layer empty capsule shell of the Intestinal flora capsule, which is made of titanium dioxide and iron oxide yellow. It is non-toxic and has the same appearance as the authentic Intestinal flora capsule.
  Other Names: Placebo control
  Arms: Placebo group

SUMMARY:
This is a single-center trial, randomized, single-blind, placebo-controlled clinical intervention study which intends to explore the safety and effectiveness of FMT capsule for the treatment of ulcerative colitis with depression.

DETAILED DESCRIPTION:
A total of 54 patients with definite diagnosis of ulcerative colitis (light-to-moderate active period) with depressive state were included. According to the random table, patients were randomly divided into the FMT capsule group and the placebo group, and received the FMT capsule and placebo interventions once a week for 4 consecutive times, respectively. The patients were followed up at the 4th, 8th and 12th week of intervention, and a simple physical examination was performed to evaluate the patient's condition changes (abdominal pain degree score, diarrhea frequency, stool characteristics and extraintestinal manifestations such as skin and joints) and modified Mayo score , IBD-QOL scale, PHQ9, SDS, HADS, HAMA, HAMD scale, etc. The improvement and effective colonization of the intestinal flora in the FMT capsule group or the placebo group of patients with depression and IBD were observed by methods such as 16S rRNA analysis of the intestinal flora In the 12th weeks.

ELIGIBILITY:
Inclusion Criteria:

1. The course of the disease is more than 6 months, and it is clearly diagnosed as ulcerative colitis with depression.【Diagnostic criteria: (2020) "JSGE Evidence-based Clinical Practice Guidelines: Inflammatory Bowel Disease" and "Chinese Mental Disorders Classification and Diagnostic Standards" (CCMD) -3) The relevant standards in the above, and also meet the improved Mayo score ≤ 10 points, PHQ9 score ≥ 5 points】;
2. There is no restriction on men and women, aged between 18-65 years old;
3. BMI is between 18-30kg/m2;
4. Have basic reading comprehension skills;
5. No other serious diseases such as heart, brain, lung, liver, and kidney are complicated;
6. Have not traveled abroad in the past month, and have no history of alcoholism, drug abuse, or smelting;
7. No antibiotics and probiotic preparations have been used within one month;
8. Agree to participate in this study and sign an informed consent form.

Exclusion Criteria:

1. Age <18 years old or >65 years old;
2. Patients with unspecified ulcerative colitis;
3. Authors with bipolar disorder, persistent mood disorder, and mania;
4. Malignant tumors such as gastrointestinal infection, irritable bowel syndrome, bowel cancer and other gastrointestinal diseases;
5. A history of gastrointestinal surgery;
6. Patients during pregnancy and lactation;
7. Complicated with obesity, hypertension, diabetes, heart disease, stroke and other serious chronic diseases (hereditary, metabolic, endocrine diseases);
8. Infectious diseases: hepatitis B or C, HIV, syphilis (rapid recovery of positive plasma), Epstein-Barr virus and cytomegalovirus infection (IgM positive);
9. Abnormal liver function: AST or ALT higher than 2 times the upper limit of normal; renal insufficiency: serum Cr higher than 1.5 times the upper limit of normal or eGFR<60ml/min; dyslipidemia (TC> 4.0 mmol/L, TG >2.0 mmol/L, LDL-c>2.5 mmol/L, HDL-c<1.0 mmol/L), CRP>8mg/L;
10. Anticoagulation therapy;
11. Patients who were participating in other clinical trials at the time of enrollment;
12. Those who do not agree to join the group or have various factors affecting compliance and other people who are not suitable for participating in clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-09-10 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 score | 12 Weeks after treatment.
  Patien Health Questionnare.The total score is 0-27 points, 0-4 points: no depression; 5-9 points: mild depression; 10-14 points: moderate depression; 15-27 points: severe depression. The higher the score, the worse the depression.

SECONDARY OUTCOMES:
SDS-score | 12 Weeks after treatment.
  Self-Rating Depression Scale.Standard total score: normal <53 points; 53-62 for mild depression; 63-72 for moderate depression; >72 for severe depression.The higher the score, the worse the depression.
HAMA-score | 12 Weeks after treatment.
  Hamilton Anxiety Scale.The total score is 0-56, among which, physical anxiety: 7-13 items; mental anxiety: 1-6 and 14 items.The higher the score, the greater the anxiety.
HAMD-score | 12 Weeks after treatment.
  Hamilton Depression Scale.The total score is 0-35 points: >35 points: severe depression; >20 points: mild or moderate depression; 8-20 may have depression; <8 points: no depression. The higher the score, the greater the depression.
HADS-score | 12 Weeks after treatment.
  Hospital Anxiety and Depression Scale.It consists of 14 (7 anxiety and 7 depression-related) scoring items, all ranging from 0-21. The higher the score, the more severe the anxiety and depression.
GSRS-score | 12 Weeks after treatment.
  Gastrointestinal Symptom Rating Scale . The score varies from 1 6 to 1 1 2 . Higher scores suggest more severe gastrointestinal pathology .
Modified Mayo score | 12 Weeks after treatment.
  Modified Mayo score for ulcerative colitis: a total of 0-12 points, scores ≤ 2 points and no single sub-item score> 1 points to clinical remission, 3 to 5 points to mild activity, 6 to 10 points to moderate activity, 11 ~12 is divided into heavy activity.The higher the score, the more severe the condition.
IBD-QoL | 12 Weeks after treatment.
  Quality of Life Analysis Table for Patients with Inflammatory Bowel Disease: There are 32 questions in total. Each question has a different level of answer from 1 to 7, 1 generation The table has the heaviest degree, and 7 represents the least degree.Total score 0-224,The higher the score, the higher the quality of life.

OTHER OUTCOMES:
WBC | 12 Weeks after treatment.
  leukocyte
CRP | 12 Weeks after treatment.
  C-reactive protein
ESR | 12 Weeks after treatment.
  erythrocyte sedimentation rate
PCT | 12 Weeks after treatment.
  procalcitonin
IL-6 | 12 Weeks after treatment.
  interleukin-6
Intestinal flora | 12 Weeks after treatment.
  16S rRNA sequencing analysis and metagenomics analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Y Ling, Principal Investigator — Army Medical Center
Locations (1):
- Department of Gastroenterology, Research Institute of Surgery, Da ping Hospital, The Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No